CLINICAL TRIAL: NCT05150977
Title: Idiopathic Hypersomnia - a Retrospective Characterization Study
Brief Title: Idiopathic Hypersomnia
Acronym: IDAHO
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-03458
Record Dates: First submitted 2021-11-26; First posted 2021-12-09 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Hypersomnia, Idiopathic
MeSH Terms: conditions — Idiopathic Hypersomnia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Idiopathic hypersomnia: Observation
  Interventions: Other: Polysomnography

INTERVENTIONS:
Other: Polysomnography — Reviewing collected data
  Other Names: Multiple sleep latency test; Questionnaires; Register data

SUMMARY:
Idiopathic hypersomnia (IH) is characterized by non-restoring night-time sleep, excessive daytime sleepiness, sleep inertia, impaired cognitive functioning and autonomic symptoms. IH seems to be long lasting, once established, but little is known about long-time consequences, and research on the relationship between idiopathic hypersomnia and all-cause mortality is however sparse. IH is thus a poorly characterized disorder of hypersomnolence, and the present study aims to answer the following research questions:

1. Are there subgroups within the IH-group, that can be retrospectively characterized out of data from polysomnography, PSG and MSLT.
2. What are the relationships between IH, and possible IH subgroups, and morbidity, mortality, and sick leave, using retrospective register data?
3. What is the natural course of IH, and possible IH subgroups, assessed with questionnaires that measures daytime sleepiness, depression, and insomnia?
4. How do subjects diagnosed with IH think about their disease, cope with it, and perceive the effects of treatments, using qualitative interviews? 185 individuals assessed and diagnosed at the Sleep unit, Uppsala university hospital between 2010-01-01 and 2019-12-31 will be contacted. After collecting informed consents, PSG and MSLT data will be analysed together with register data regarding morbidity, mortality, sick leave, and pharmacotherapy.Questionnaires used at the time of the original assessment will be reviewed and, to study the natural course of the syndrome, the same questionnaires will be sent to the participants by mail.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic hypersomnia, according to the The International Classification of Sleep Disorders - Third Edition (ICSD-3)

Exclusion Criteria:

* Other serious somatic or psychiatric disease
* Drug additction with drug seeking behaviour

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible subjects are 185 individuals with idiopathic hypersomnia (IH) assessed and diagnosed using polysomnography and multiple sleep latency test at the Sleep unit, Uppsala university hospital between 2010-01-01 and 2019-12-31. Inclusion criteria is IH, according to the ICSD-3.
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Polysomnography | Baseline
  Spectral analyses
Multiple sleep latency test | Baseline
  Sleep latency and REM latency

SECONDARY OUTCOMES:
Morbidity | 1 week
  Diagnoses
Sick leave | 1 week
  Percent
Pharmacotherapy | 1 week
  Type and dosage
Epworth Sleepiness Scale | Baseline
  Score on a scale with a total score of 0 to 24. Higher values means more severe problems.
Sleep Problem Acceptance Questionnaire | 1 week
  Score on a scale. An 8-item self-report questionnaire, total scores range from 0 to 48 points. Higher values equals higher level of acceptance and a positive outcome.
Insomnia Severity Index | Baseline
  Score on a scale. Seven items with a total score ranging from 0 to 28 points. Higher values means more severe insomnia, a negative outcome.
Montgomery Åsberg Depression Rating Scale | Baseline
  Score on a scale. Higher score indicates more severe depression, a negative outcome. The overall score ranges from 0 to 60.
Diurnal Type Questionnaire | Baseline
  Score on a scale. The overall score ranges 0 to 21, and higher scores equals more of a delayed sleep phase.
Munich Parasomnia Screening | Baseline
  Score on a scale. 21 items with an overall score ranging from 0 to 84. Higher scores indicates a negative outcome.
The Ullanlinna Narcolepsy Scale | Baseline
  Score on a scale. 11 item with a total score ranging 0-44. Higher total score equals a negative outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Karlsten, PhD, Study Chair — Uppsala University
Locations (1):
- Uppsala University, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Undecided